CLINICAL TRIAL: NCT03844139
Title: Observation of Effect and Complication of Two Types of Nasogastric Tube Feeding Enteral Nutrition for Elderly Dysphagia Patients After Stroke
Brief Title: Effect and Complication of Two Types of Nasogastric Tube Feeding for Elderly Dysphagia Patient After Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: zhang yuejiao
Record Dates: First submitted 2019-02-01; First posted 2019-02-18 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Feeding pump group(continous): Using the feeding pump to give patients prescribed enteral nutrient solution through nasogastric tube in 24 hours
  Interventions: Device: Feeding pump and glycerin syringe
- Glycerin syringe group(intermittent): Using the glycerin syringe to give patients prescribed enteral nutrient solution through nasogastric tube in 4-5 times
  Interventions: Device: Feeding pump and glycerin syringe

INTERVENTIONS:
Device: Feeding pump and glycerin syringe — The continuous group use feeding pump and the intermittent group use syringe to give dysphagia patients after stroke prescribed nutrition through nasogastric tube.

SUMMARY:
Dysphagia is a common problem after stroke.Patients after stroke with swallow problem will have a nasogastric tube to be feeded. In this study , investigators have including and excluding criteria. Continous feeding group and intermittent feeding group had been widely used in enteral nutrition feeding in investigators' institution. Investigators will observe participants' nutrition condition and tube-feeding related complications. In continous group patients, participants usually are given prescribed enteral nutrient solution using nutrition pump in 24 hours; while in intermittent feeding group, participants will be given prescribed enteral nutrient solution in 4-5 times by special syringe. During the whole process, investigators will observe all participants' nutrition condition (body mass index, plasma albumin and calf girth) and tube-feeding related complications( regurgitation, aspiration,gastric retention, diarrhea,constipation). With all those data, the investigators will assess which feeding type is better.

ELIGIBILITY:
Inclusion Criteria:

* Older than 65 years old
* Clinical diagnosis of stroke( ischemic and hemorrhage)
* With moderate and/or sever swallow problem(water swallow test IV-V degree)
* With nasogastric feeding tube more than 4 weeks
* Do rehabilitation in our hospital or designated hospitals

Exclusion Criteria:

* Without nasogastric feeding tube
* Patients with fever and other infection
* Chronic or acute anoxia
* Poor obedience
* Quit treatment or go back home to take rehabilitation
* Critically ill or died

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Every 50 patients in each group
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-13 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
weight | 4-6 weeks
  weight in kilogram every week
plasma albumin | 4-6 weeks
  plasma albumin every week
tube-feeding related complications( regurgitation, aspiration,gastric retention, diarrhea,constipation) | 4-6 weeks
  incidence of each complication

SECONDARY OUTCOMES:
calf girth | 4-6 weeks
  length of calf girth

CONTACTS AND LOCATIONS:
Locations (1):
- Zhangy Yuejiao, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No